CLINICAL TRIAL: NCT01117740
Title: Comparative Effectiveness of Indwelling Pleural Catheters Versus Thoracoscopic Pleurodesis for Treatment of Malignant Pleural Effusions
Brief Title: Pleural Catheters Versus Thoracoscopic Pleurodesis
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0103
Record Dates: First submitted 2010-04-20; First posted 2010-05-05 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Lung Cancer
Keywords: Malignant Pleural Effusions; MPE; Lungs; Quality of Life; M. D. Anderson Symptom Inventory; MDASI; Indwelling Pleural Catheters; Thoracoscopic Pleurodesis; Symptom burden; Pleurodesis efficacy; Complications; Health care resource utilization
MeSH Terms: conditions — Lung Neoplasms; Pleural Effusion, Malignant | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thoracoscopy Group
  Interventions: Behavioral: MDASI Questionnaire
- Indwelling Pleural Catheters
  Interventions: Behavioral: MDASI Questionnaire

INTERVENTIONS:
Behavioral: MDASI Questionnaire — 19 question M. D. Anderson Symptom Inventory (MDASI) before pleural effusion treatment and at each follow-up visit, takes about 5 minutes to complete each time.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to compare 2 different methods for treating a pleural effusion. Researchers also want to learn how the treatment you receive effects your quality of life (your ability to do the things you like to do and how happy you feel.

DETAILED DESCRIPTION:
If you agree to take part in this study, you may be asked to fill out a questionnaire called the MD Anderson Symptom Inventory (MDASI) before your scheduled pleural effusion treatment procedure, 24 hours after your procedure, and then weekly for the next 4 months. During this time, a member of the study staff or a computer system will call you at home on your desired day and time to complete the questionnaire. The MDASI for lung-related symptoms has 22 questions about the possible symptoms caused by the disease, and how the symptoms may affect the activities of your daily life, which you will rate on a scale of 0-10. The MDASI will take about 5 minutes to complete each time.

You will also complete 2 questionnaires called the SF6D Patient Self Assessment and Borg Scale before your scheduled pleural effusion treatment procedure, 2 weeks later, and then 1 time a month for 1 year. These questionnaires are part of your standard of care. There are 7 questions total about how the symptoms may affect the activities of your daily life. If you are not in the clinic, a member of the study staff will call you at home on your desired day and time to complete the questionnaires. The questionnaires should take about 5 minutes total to complete each time.

Your information will be stored in a password-protected database for use in future research related to cancer for up to 5 years after the study is completed.

Before any of your information that is stored in the database can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of MD Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at MD Anderson, including research involving your data from this bank, must first be approved by the IRB.

Your information will be given a code number so that none of your personal identifying information will be directly linked to your information. Only the researcher in charge of the database will have access to the code numbers and be able to link the information in the database back to you. Other researchers who use the database will not be able to link your information or file back to you.

This is an investigational study. Up to 445 participants will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MPE who are suitable for either pleural catheter placement or thoracoscopic pleurodesis who subsequently have either procedure performed
2. Sufficient mental capacity to answer SF-6D and Borg score questions
3. Age 18 or older
4. Life expectancy > 2 months
5. English or Spanish speaking

Exclusion Criteria:

1. Patients undergoing pleurodesis for benign disease (e.g., spontaneous pneumothorax)
2. Inability or unwillingness to give informed consent
3. Inability to perform phone call follow-up
4. Pregnancy
5. Previous intrapleural therapy for MPE
6. Prior radiation therapy encompassing the entire hemithorax
7. Chylous effusions associated with malignant disease
8. Bilateral effusions requiring bilateral pleurodesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, 18 years or older, with malignant pleural effusions, suitable for either pleural catheter placement or thoracoscopic pleurodesis.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2010-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quality-Adjusted Survival Times | 12 Months with follow up until death or recurrence
  Quality-adjusted time to death (measured as QALYs) for two patient groups (indwelling pleural catheters and thoracoscopy), calculated using Brazier's SF-6D utility measure described to determine utilities, then integrating utilities over time to arrive at quality-adjusted survival for each patient.

SECONDARY OUTCOMES:
Patient Responses to MDASI | Monthly beginning at pleural effusion treatment
  M. D. Anderson Symptom Inventory (MDASI) symptoms questionnaire: 19 questions about symptoms rated on a scale of 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: David Ost, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ost DE, Jimenez CA, Lei X, Cantor SB, Grosu HB, Lazarus DR, Faiz SA, Bashoura L, Shannon VR, Balachandran D, Noor L, Hashmi YB, Casal RF, Morice RC, Eapen GA. Quality-adjusted survival following treatment of malignant pleural effusions with indwelling pleural catheters. Chest. 2014 Jun;145(6):1347-1356. doi: 10.1378/chest.13-1908. PMID 24480929
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org